CLINICAL TRIAL: NCT07144033
Title: Butyrate and Taurine for Chronic Postsurgical Pain in Adult Cardiac Surgical Patients: Bayesian Optimized Double-blinded Randomized Controlled Trial
Brief Title: Butyrate and Taurine for Chronic Postsurgical Pain in Adult Cardiac Surgical Patients
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, WONG MAN KIN, Assistant Professor, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2025.335-T
Record Dates: First submitted 2025-08-20; First posted 2025-08-27 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-08

CONDITIONS: Pain, Acute; Pain, Chronic; Chronic Post Operative Pain
MeSH Terms: conditions — Acute Pain; Chronic Pain; Pain, Postoperative | interventions — Butyrates; Taurine

STUDY DESIGN:
Intervention Model Description: double-blinded, randomized, placebo-controlled trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Patients are randomly allocated to combined taurine/butyrate or identical-looking capsules by drawing sequentially numbered, coded, sealed, opaque envelops, each containing the type of intervention assignment or placebo. The sealed envelopes for randomization are prepared by a third party who took no further part in the study. The study investigators, the primary care team and the participants are masked to the group assignments. This is achieved by using an indistinguishable placebo (a proprietary product from Colorcon called StarCap - a mixture of Pregelatinized Maize Starch and Maize Starch) capsules manufactured by an independent pharmaceutical company in Western Australia.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- butyrate/taurine group (Experimental): Interventional group (combination of taurine and butyrate): 4g of taurine plus 4.8g of sodium butyrate will be administered orally after enrolment on the day before surgery, and then daily thereafter for three months after surgery.
  Interventions: Dietary Supplement: Butyrate and Taurine
- Placebo control (Placebo Comparator): Placebo group: indistinguishable placebo capsules will be administered orally after enrolment on the day before surgery, followed by daily administration for three months after surgery. Both taurine, butyrate and the indistinguishable placebo capsules are white in color.
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Butyrate and Taurine — This dose of butyrate is chosen to maximize any treatment effect in postoperative pain. Butyrate was reported to be safe at this dose for a prolonged period of 8 weeks. The dose of taurine is considered safe according to the European Food Safety Authority and was used in previous human perioperative trials. A human pharmacokinetic study showed that after taking 4g taurine (32 mmol) orally, plasma taurine levels reached a peak level of 86 mg/L (or 0.7 mmol/L) at 1.5 hours, exceeding the physiological plasma taurine level (0.01-0.1 mmol/L), which is needed to exert its pharmacological benefits.
  Arms: butyrate/taurine group
Other: Placebo — indistinguishable placebo capsules will be administered orally after enrolment on the day before surgery, followed by daily administration for three months after surgery.
  Arms: Placebo control

SUMMARY:
This study is a single-center, phase II, randomized, placebo-controlled, Bayesian-designed, double-blinded trial

Goal and Questions:

The primary goal is to evaluate if a combination of taurine and butyrate can reduce chronic postsurgical pain (CPSP) in adult cardiac surgical patients. The study also aims to determine if these compounds are safe, effective in perioperative pain control, and feasible for improving postoperative outcomes.

Participants:

The study will include adult patients (aged 18 or older) undergoing elective coronary artery bypass graft (CABG), valve repair/replacement, combined CABG/valve, or major aortic procedure via sternotomy. Exclusion criteria include emergency surgery, redo surgery, a history of chronic pain or chronic opioid/sedative use, and an estimated glomerular filtration rate (eGFR) less than 30 mL/min. The target sample size is 216 patients.

Intervention group: Patients will receive 4g of taurine and 4.8g of sodium butyrate orally once daily, starting the day before surgery and continuing for three months post-surgery.

Placebo group: Patients will receive indistinguishable placebo capsules orally once daily, following the same schedule as the intervention group.

Primary Outcome: The incidence of chronic postsurgical pain at 3 months,

Secondary Outcomes:

Quality of Recovery Questionnaire (QoR-15) at 72 hours after extubation.

Pain scores (NRS) at rest and with movement at 12, 24, 48, and 72 hours post-extubation.

Postoperative morphine requirements and time to first morphine rescue.

Incidence of opioid-related side effects, such as postoperative nausea and vomiting (PONV).

Duration of mechanical ventilation, and length of stay in the ICU and hospital.

Long-term pain assessment using the Short-Form McGill Pain Questionnaire-2 (SF-MPQ-2), Brief Pain Inventory (BPI) Interference Scale, and Neuropathic Pain Questionnaire (NPQ) at 1, 3, 6, and 12 months post-surgery

Proteomic analysis:

Blood samples within 72 hours after surgery will be collected for proteomic analysis to investigate predictors for chronic postsurgical pain.

DETAILED DESCRIPTION:
INTRODUCTION

Managing pain after cardiac surgery is a complex challenge. Traditional pain medications like opioids and NSAIDs are effective but come with significant side effects, including addiction, respiratory issues, and organ damage. This has led researchers to look for safer alternatives. Two promising compounds are butyrate and taurine. Butyrate is a short-chain fatty acid produced by gut bacteria. It helps reduce inflammation and pain by influencing both the central and peripheral nervous systems. Studies show that it can alleviate various types of pain, from visceral to neuropathic, and may help prevent chronic pain after surgery. Taurine is an amino acid that modulates neurotransmitters and ion channels in the nervous system, providing an analgesic effect. It may also reduce opioid tolerance, which is crucial for managing long-term pain. The innovative approach of this research is to use both butyrate and taurine together. Butyrate's anti-inflammatory properties complement taurine's pain-modulating effects, creating a synergistic combination. This could not only reduce the need for traditional opioids-thus minimizing their side effects-but also improve the overall quality of recovery for cardiac surgery patients. Both compounds are safe, cost-effective, and readily available as oral supplements, making them a practical and viable alternative for modern pain management.

METHODS AND ANALYSIS

Study population and design This is a single-centre, phase II, randomized, placebo-controlled, Bayesian designed double-blinded trial conducted at Prince of Wales Hospital, a tertiary hospital in Hong Kong.

Randomization and Concealment Patients are randomly allocated to combined taurine/butyrate or identical-looking capsules by drawing sequentially numbered, coded, sealed, opaque envelops, each containing the type of intervention assignment or placebo. The sealed envelopes for randomization are prepared by a third party who took no further part in the study. The study investigators, the primary care team and the participants are masked to the group assignments. This is achieved by using an indistinguishable placebo (a proprietary product from Colorcon called StarCap - a mixture of Pregelatinized Maize Starch and Maize Starch) capsules manufactured by an independent pharmaceutical company in Western Australia.

Blood sampling Animal models suggested a positive correlation of serum butyrate concentration on T-cell function for treatment responsive cancer patients in the range of 0.1-0.2 mcg/ml, and an inverse relationship of a similar serum concentration in treatment response in schizophrenic patients. However, the plasma level that is required for analgesia in humans has not yet been established. To ensure the study drugs reach a clinically meaningful plasma concentration after gut absorption and hepatic first-pass, blood samples will be collected within 72-hour after surgery to analyse taurine and butyrate levels.

Since postoperative inflammation peaks at 12-24 hours and declines to normal at 48-72 hours in the absence of complications, blood samples within 72-hour after surgery will be collected for proteomic analysis. By integrating proteomic data with perioperative clinical variables, predictors for chronic postsurgical pain, as well as modifiable factors that influence pain outcomes can be identified.

Compliance check Drug compliance will be check via blood sampling and rectal swab. Plasma levels of taurine and butyrate will be measured at baseline after taking informed consent, and at 1 and 3 months after surgery. Similarly, rectal swab for butyrate and taurine level will be measured at the same time points. Rectal swab is performed by the research nurse. Since the study drug capsules will all be given to the participants before post-surgical hospital discharge, the number of remaining capsules will be counted during follow-up visits to check for the compliance.

Statistical Analysis The study adopts a Bayesian framework to evaluate the efficacy of a novel combination of butyrate and taurine in reducing the incidence of CPSP at 3 months. A sample size of 180 patients (90 per arm) based on Bayesian simulation (Department of Biostatistics, The University of Texas MD Anderson Cancer Centre, https://biostatistics.mdanderson.org/shinyapps/rBOP2/) indicates a power 87.0% to detect an absolute risk reduction in chronic pain incidence of 20% (from a baseline of 30% to 10%). The clinically meaningful absolute risk reduction in CPSP is set at 6%. Should non-futility be demonstrated in this phase II trial, it will provide baseline data to inform future research for demonstration on superiority.

Considering a drop-out of 20%, the overall sample size is increased to 216 patients (108 per arm). Blinded interim analyses will be conducted at every 72 randomized patients until the target sample size 216 are randomized. The conditions for stopping for superiority and futility are as follows:

* Stopping for Efficacy: If the posterior probability of a clinically meaningful reduction in CPSP (≥6%) exceeds 95%, the trial will stop, and the combination of butyrate and taurine will be deemed effective.
* Stopping for futility: If the posterior probability of achieving a meaningful reduction in CPSP incidence is less than 5%, the trial will stop and the intervention will be considered ineffective. A demonstrated non-futility can provide baseline data to inform future larger-scale trials with adequate power to demonstrate superiority.
* Continuing to the next stage: If the posterior probability lies between 5% and 95%, the trial will proceed to the next interim analysis, and an additional 66 patients (33 per group) will be recruited.

Analysis of Posterior Probabilities

At each stage, the posterior probability of achieving a ≥6% reduction in CPSP incidence will be calculated using the Bayesian hierarchical model as described above. The posterior distribution of the effect size will be summarized by:

* The posterior mean and 95% credible intervals for the reduction in CPSP incidence
* The posterior probability of achieving the predicted minimum clinically important difference (MCID) of 6%.

Continuous outcomes will be analyzed using Bayesian hierarchical models and reported as mean (standard deviation) or median (interquartile range) as appropriate after checking for normality using the Shapiro-Wilk's test. Categorical outcomes will be compared with Chi-square test. Generalized Estimating Equations (GEE) models will be conducted to evaluate the analgesia time effects between group. SPSS 27.0 (IBM Corp, Armonk, NY) is used for data analyses and Stata V.14 (Stata, College Station, Texas, USA) is used to conduct GEE with a Gaussian distribution, identity-link function, exchangeable correlation with robust standard error (SE). Level of significance will be set at P<0.05 without adjusting for multiple comparisons.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients aged 18 or older
* elective surgery
* coronary artery bypass graft (CABG), valve repair/replacement, combined CABG/valve procedure, or major aortic procedure via sternotomy

Exclusion Criteria:

* emergency surgery
* redo surgery
* history of chronic pain or on chronic opioids/sedatives
* already taking taurine or butyrate prior to enrolment
* renal failure with estimated glomerular filtration rate <30mL/min (calculated by Cockcroft-Gault formula)
* re-operation within 24 hours after surgery
* intraoperative use of remifentanil
* inability to provide informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 216 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2027-01-31 (Estimated); Study Completion 2028-01-31 (Estimated)

PRIMARY OUTCOMES:
Chronic postsurgical pain at 3 months | At 3 months after surgery
  Incidence of chronic postsurgical pain based on the IASP definition

SECONDARY OUTCOMES:
chronic postsurgical pain at 1 month | At 1 month after surgery
  Incidence of chronic postsurgical pain based on IASP definition
chronic postsurgical pain at 6 month | At 6 months after surgery
  Incidence of chronic postsurgical pain based on IASP definition
chronic postsurgical pain at 12 month | At 12 months after surgery
  Incidence of chronic postsurgical pain based on IASP definition
Brief Pain Inventory (BPI) at 1 month | At 1 month after surgery
  The functional and affective interference of chronic postsurgical pain: the pain score is scaled from 0-10, the higher the score, the worse the pain. The functional and affective interference scale ranges from 0-10, the lower the score, the worse the performance
Brief Pain Inventory (BPI) at 3 month | At 3 month after surgery
  The functional and affective interference of chronic postsurgical pain: the pain score is scaled from 0-10, the higher the score, the worse the pain. The functional and affective interference scale ranges from 0-10, the lower the score, the worse the performance
Brief Pain Inventory (BPI) at 6 month | At 6 month after surgery
  The functional and affective interference of chronic postsurgical pain: the pain score is scaled from 0-10, the higher the score, the worse the pain. The functional and affective interference scale ranges from 0-10, the lower the score, the worse the performance
Brief Pain Inventory (BPI) at 12 month | At 12 month after surgery
  The functional and affective interference of chronic postsurgical pain: the pain score is scaled from 0-10, the higher the score, the worse the pain. The functional and affective interference scale ranges from 0-10, the lower the score, the worse the performance
Neuropathic Pain Questionnaire (NPQ) at 1 month | At 1 month after surgery
  To detect the presence of severity of neuropathic pain. The scale ranges from 0-100. The higher the score, the worse the neuropathic pain
Neuropathic Pain Questionnaire (NPQ) at 3 month | At 3 month after surgery
  To detect the presence of severity of neuropathic pain. The scale ranges from 0-100. The higher the score, the worse the neuropathic pain
Neuropathic Pain Questionnaire (NPQ) at 6 month | At 6 month after surgery
  To detect the presence of severity of neuropathic pain. The scale ranges from 0-100. The higher the score, the worse the neuropathic pain
Neuropathic Pain Questionnaire (NPQ) at 12 month | At 12 month after surgery
  To detect the presence of severity of neuropathic pain. The scale ranges from 0-100. The higher the score, the worse the neuropathic pain
Short-Form McGill Pain Questionnaire-2 (SF-MPQ-2) at 1 month | At 1 month after surgery
  To determine the functional and affective interference of chronic pain. 22-item questionnaire ranges from 0-100. The higher the score, the worse the pain interference
Short-Form McGill Pain Questionnaire-2 (SF-MPQ-2) at 3 month | At 3 month after surgery
  To determine the functional and affective interference of chronic pain. 22-item questionnaire ranges from 0-100. The higher the score, the worse the pain interference
Short-Form McGill Pain Questionnaire-2 (SF-MPQ-2) at 6 month | At 6 month after surgery
  To determine the functional and affective interference of chronic pain. 22-item questionnaire ranges from 0-100. The higher the score, the worse the pain interference
Short-Form McGill Pain Questionnaire-2 (SF-MPQ-2) at 12 month | At 12 month after surgery
  To determine the functional and affective interference of chronic pain. 22-item questionnaire ranges from 0-100. The higher the score, the worse the pain interference
Quality of Recovery Questionnaire (QoR-15) | At 72 hours after extubation
  15-item questionnaire to determine to quality of recovery. Each item score ranges from 0-10. The higher the score, the worse the condition.
Numerical Rating Scale (NRS) pain scores at rest at 12h | At 12 hours after extubation
  Pain score at rest. It ranges from 0-10. The higher the score, the worse the pain
Numerical Rating Scale (NRS) pain scores at rest at 24h | At 24 hours after extubation
  Pain score at rest. It ranges from 0-10. The higher the score, the worse the pain
Numerical Rating Scale (NRS) pain scores at rest at 48h | At 48 hours after extubation
  Pain score at rest. It ranges from 0-10. The higher the score, the worse the pain
Numerical Rating Scale (NRS) pain scores at rest at 72h | At 72 hours after extubation
  Pain score at rest. It ranges from 0-10. The higher the score, the worse the pain
Numerical Rating Scale (NRS) pain scores at movement at 12h | At 12 hours after extubation
  Pain score at movement. Maximal pain score according to patient. It ranges from 0-10. The higher the score, the worse the pain.
Numerical Rating Scale (NRS) pain scores at movement at 24h | At 24 hours after extubation
  Pain score at movement. Maximal pain score according to patient. It ranges from 0-10. The higher the score, the worse the pain.
Numerical Rating Scale (NRS) pain scores at movement at 48h | At 48 hours after extubation
  Pain score at movement. Maximal pain score according to patient. It ranges from 0-10. The higher the score, the worse the pain.
Numerical Rating Scale (NRS) pain scores at movement at 72h | At 72 hours after extubation
  Pain score at movement. Maximal pain score according to patient. It ranges from 0-10. The higher the score, the worse the pain.
Patient-controlled analgesia machine morphine consumption at 12h | At 12 hours after extubation
  Postoperative morphine requirement based on patient-controlled analgesia machine
Patient-controlled analgesia machine morphine consumption at 12h | At 24 hours after extubation
  Postoperative morphine requirement based on patient-controlled analgesia machine
Patient-controlled analgesia machine morphine consumption at 12h | At 48 hours after extubation
  Postoperative morphine requirement based on patient-controlled analgesia
Patient-controlled analgesia machine morphine consumption at 12h | At 72 hours after extubation
  Postoperative morphine requirement based on patient-controlled analgesia
Time for the first dose of morphine as recorded on patient-controlled analgesia machine | Within 48 hours after surgery
  The time of first requirement of postoperative morphine based on patient-controlled analgesia
Time weaned to spontaneous breathing | within 48 hours after surgery
  Time weaned to spontaneous breathing based on the ASV ventilator protocol
Exutubation time | within 72 hours after surgery
  Time of extubation after surgery
Patient satisfaction to pain management at 12 hours | At 12 hours after surgery
  Patient satisfaction to pain management on scale 0-100
Patient satisfaction to pain management at 24 hours | At 24 hours after surgery
  Patient satisfaction to pain management on scale 0-100
Patient satisfaction to pain management at 48 hours | At 48 hours after surgery
  Patient satisfaction to pain management on scale 0-100
Patient satisfaction to pain management at 72 hours | At 72 hours after surgery
  Patient satisfaction to pain management on scale 0-100
Postoperative nausea or vomiting | Within 72 hours after surgery
  Number of episodes of postoperative nausea or vomiting
Oral analgesic use | Within 72 hours after surgery
  Prescription and the number of additional analgesics after surgery
surgical site infection | Within 30 days after surgery
  Surgical site infection based on standard CDC definition
Length of stay in ICU | Within 1 week after surgery
  Number of days spent in ICU
Length of stay in hospital | Within 30 days after surgery
  Number of days spent in hospital
Proteomics analysis | Within 72 hours after surgery
  Blood sampling for proteomics at 48-72 hours afters surgery

CONTACTS AND LOCATIONS:
Overall Officials: Henry Wong, MBChB, Principal Investigator — Department of Anaesthesia and Intensive Care, The Chinese University of Hong Hong
Locations (1):
- Prince of Wales Hospital, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: Yes
The principal investigator has to be contacted for sharing of IPD information
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: Within 5 years upon completion of the study
Access Criteria: The principal investigator of the study has to be informed for access right of the study information